CLINICAL TRIAL: NCT00489541
Title: A Prospective Evaluation in a Non-Randomized Trial of the Safety and Efficacy of the Use of the TAXUS® ElementTM Paclitaxel-Eluting Coronary Stent System for the Treatment of De Novo Coronary Artery Lesions in Small Vessels
Brief Title: TAXUS PERSEUS Small Vessel
Acronym: PERSEUS SV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2043; S2043-PIVOT-2006
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Results first posted 2011-06-28 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Artery Disease
Keywords: paclitaxel-eluting stent; PES
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TAXUS Element Stent System (Experimental)
  Interventions: Device: Percutaneous Coronary Intervention (PCI) with paclitaxel-eluting stent (TAXUS Element) implantation

INTERVENTIONS:
Device: Percutaneous Coronary Intervention (PCI) with paclitaxel-eluting stent (TAXUS Element) implantation — TAXUS Element stent implantation

SUMMARY:
The purpose of the TAXUS PERSEUS Small Vessel trial is to evaluate the safety and efficacy of the next-generation Boston Scientific TAXUS paclitaxel-eluting coronary stent system (TAXUS® ElementTM) for the treatment of de novo atherosclerotic lesions of up to 20 mm in length in native coronary arteries of ≥ 2.25 mm to < 2.75 mm diameter.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm superiority trial to assess the TAXUS® Element™ Paclitaxel-Eluting Coronary Stent System for the treatment of de novo atherosclerotic lesions of ≤20 mm in length in native coronary arteries with visual RVD of ≥ 2.25 mm to < 2.75 mm diameter.

Two hundred twenty-four (224) subjects will be treated with the TAXUS Element stent at a maximum of 35 clinical sites. Follow-up at 30 days, 9 months including angiography) and 1 year will be completed in all subjects enrolled in the study. Eligible subjects will have annual follow-up until 5 years post-index procedure.

ELIGIBILITY:
Clinical Inclusion Criteria:

* Subject is ≥ 18 years old
* Eligible for percutaneous coronary intervention (PCI)
* Documented stable angina pectoris (Canadian Cardiovascular Society [CCS] Classification 1, 2, 3, or 4) or unstable angina pectoris (Braunwald Class IB-C, IIB-C, or IIIB-C), or documented silent ischemia
* Acceptable candidate for coronary artery bypass grafting (CABG)
* Left ventricular ejection fraction (LVEF) is ≥ 30%
* Subject (or legal guardian) understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
* Subject willing to comply with all specified follow-up evaluations

Clinical Exclusion Criteria:

* Contraindication to aspirin (ASA), or to both clopidogrel and ticlopidine
* Known hypersensitivity to paclitaxel
* Known allergy to stainless steel
* Known allergy to platinum
* Previous treatment of the target vessel with any anti-restenotic drug-coated or drug-eluting coronary stent
* Previous treatment of the target vessel with a bare metal stent (BMS) within 9 months of the index procedure
* Previous treatment of any non-target vessel with any anti-restenotic drug-coated or drug-eluting coronary stent within 9 months of the index procedure
* Previous treatment with intravascular brachytherapy in the target vessel
* Planned PCI or CABG post-index procedure
* Planned or actual target vessel treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon or transluminal extraction catheter immediately prior to stent placement
* Myocardial infarction (MI) within 72 hours prior to index procedure
* Cerebrovascular accident (CVA) within the past 6 months
* Cardiogenic shock
* Acute or chronic renal dysfunction
* Prior anaphylactic reaction to contrast agents
* Leukopenia
* Thrombocytopenia
* Thrombocytosis
* Active peptic ulcer or active gastrointestinal (GI) bleeding
* Current treatment, or past-treatment within 12-months of the index procedure, with paclitaxel or other chemotherapeutic agents
* Anticipated treatment with paclitaxel or oral rapamycin during any period in the 9-months after the index procedure
* Known intention to procreate within 9 months after the index procedure
* Positive pregnancy test within 7 days before the index procedure, or lactating
* Life expectancy of less than 24 months due to other medical conditions
* Co-morbid condition(s) that could limit subject's ability to comply with study follow-up requirements or impact study scientific integrity
* Currently participating in another investigational drug or device study

Angiographic Inclusion Criteria:

* Target Lesion

  * Target lesion located in native coronary artery
  * Target lesion must be de novo
  * Target lesion diameter stenosis ≥ 50%
  * Reference vessel diameter (RVD) ≥ 2.25 mm to < 2.75 mm
  * Cumulative target lesion length ≤ 20 mm (area to be treated may be composed of multiple lesions but must be completely coverable by one study stent)
  * Target lesion is successfully pre-dilated
* One non-target lesion may be treated in a non-target vessel as follows:

  * Non-target lesion in non-target vessel must be treated with commercially available TAXUS stent if use of drug eluting stent required
  * Treatment must be deemed a clinical angiographic success, without requiring use of unplanned additional stents(s)
  * Treatment must be completed prior to treatment of target vessel

Angiographic Exclusion Criteria:

* Target lesion located in left main artery, whether protected or unprotected
* Target lesion is a chronic total occlusion (TIMI flow ≤ 1)
* Target lesion is restenotic
* Target lesion is located in a saphenous vein graft or mammary artery graft
* Target lesion is accessed via saphenous vein graft or mammary artery graft
* Target lesion is < 5 mm from bare metal stent (BMS)
* Target lesion < 5 mm from ostium
* Target lesion < 5 mm from side branch vessel ≥ 2.0 mm in diameter (Exceptions: subject may be enrolled if side branch is 100% occluded or if side branch is protected with a patent graft)
* Untreated lesions with ≥ 50% diameter stenosis or thought to impair flow remaining in target vessel at a location with ≥ 2.0mm RVD
* Target lesion and/or target vessel proximal to target lesion moderately severely calcified
* Target lesion and/or target vessel proximal to target lesion severely tortuous
* Target lesion located within or distal to a > 60° bend in target vessel
* Target vessel with angiographic presence of probable or definite thrombus
* Unprotected left main coronary artery disease
* Protected left main coronary artery disease with target lesion in Left Anterior Descending artery (LAD) or Left Circumflex artery (LCx). Subject may be enrolled if only lesion is target lesion in Right Coronary Artery (RCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean J Kereiakes, MD, Principal Investigator — The Christ Hospital; Louis A Cannon, MD, Principal Investigator — Cardiac and Vascular Research Center of Northern Michigan
Locations (28):
- United States (28):
  - Medical Center East, Birmingham, Alabama
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Scripps Clinic, La Jolla, California
  - Christiana Hospital, Newark, Delaware
  - Mediquest Research at Munroe Regional Medical Center, Ocala, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - St. John's Hospital, Springfield, Illinois
  - Northern Indiana Research Alliance / Lutheran Hospital of Indiana, Fort Wayne, Indiana
  - Maine Medical Center, Portland, Maine
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Nebraska Heart Hospital, Lincoln, Nebraska
  - St. Joseph's Hospital Health Center, Liverpool, New York
  - Lenox Hill Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Main Line Health Heart Center, Bryn Mawr, Pennsylvania
  - Methodist DeBakey Heart Center, Houston, Texas
  - TexSAn Heart Hospital, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Derived] Allocco DJ, Cannon LA, Britt A, Heil JE, Nersesov A, Wehrenberg S, Dawkins KD, Kereiakes DJ. A prospective evaluation of the safety and efficacy of the TAXUS Element paclitaxel-eluting coronary stent system for the treatment of de novo coronary artery lesions: design and statistical methods of the PERSEUS clinical program. Trials. 2010 Jan 7;11:1. doi: 10.1186/1745-6215-11-1. PMID 20059766

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects were enrolled at 28 United States centers between July 13, 2007 and August 27, 2008. All subjects were required to undergo angiographic assessment at 9 months. The historic control group consists of 125 matched bare metal Express subjects from the TAXUS V trial (NCT00301522), including 108 with 9-month QCA follow-up.
Groups:
- TAXUS Element: Paclitaxel-eluting stent (PES) implanted using standard percutaneous coronary intervention (PCI) technique
- Historical Control Bare Metal Stent (BMS): The control group consists of 125 matched bare metal Express subjects from the TAXUS V trial (NCT00301522).
Period: 12-Month Clinical Follow-up
Arm/Group | TAXUS Element | Historical Control Bare Metal Stent (BMS)
Started | 224 | 125
Completed | 215 | 120
Not Completed | 9 | 5
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Missed 12-Month Visit | 2 | 0
Not completed — Death | 3 | 2
Period: 9-Month Angiographic Follow-up
Arm/Group | TAXUS Element | Historical Control Bare Metal Stent (BMS)
Started | 224 | 125
Completed | 197 | 108
Not Completed | 27 | 17
Not completed — No 9-Month Angiography Performed | 23 | 12
Not completed — Not Evaluable for 9-Month Angiography | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAXUS Element | Historical Control Bare Metal Stent (BMS) | Total
Number analyzed (Participants) | 224 | 125 | 349
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 63 | 163
  >=65 years | 124 | 62 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.3) | 64.2 (10.9) | 64.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 49 | 130
  Male | 143 | 76 | 219
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 11 | 3 | 14
  Caucasian | 204 | 115 | 319
  Asian | 0 | 0 | 0
  Black of African heritage | 6 | 5 | 11
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska native | 1 | 0 | 1
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 224 | 125 | 349
Cardiac History [Number; unit: participants] — The same participant may be included in more than one category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    Previous Percutaneous Coronary Intervention (PCI) | 92 | 42 | 134
    Previous Coronary Artery Bypass Graft (CABG) | 41 | 24 | 65
    Previous Myocardial Infarction (MI) | 57 | 36 | 93
    Congestive Heart Failure | 18 | 3 | 21
    Stable Angina | 136 | 70 | 206
    Unstable Angina | 45 | 37 | 82
    Silent Ischemia | 43 | 18 | 61
Cardiac History: Ejection Fraction [Mean (Standard Deviation); unit: ejection fraction percent] | 57.9 (9.4) | 55.0 (9.2) | 56.8 (9.4)
Cardiac Risk Factors [Number; unit: participants] — The same participant may be included in more than one category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    Smoking, Ever | 137 | 69 | 206
    Medically Treated Diabetes | 82 | 40 | 122
    Hyperlipidemia Requiring Medication | 191 | 97 | 288
    Hypertension Requiring Medication | 181 | 100 | 281
    Family History of Coronary Artery Disease | 144 | 73 | 217
Comorbidities [Number; unit: participants] — The same participant may be included in more than one category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Peripheral Vascular Disease | 24 | 14 | 38
    Transient Ischemic Attack/Cerebrovascular Accident | 21 | 5 | 26
    History of Renal Disease | 9 | 0 | 9
    History of Gastrointestinal Bleeding | 5 | 2 | 7
Lesion Characteristic: Target Lesion Vessel [Number; unit: participants]
  Left Anterior Descending | 85 | 53 | 138
  Left Circumflex | 93 | 45 | 138
  Right Coronary Artery | 46 | 27 | 73
Lesion Characteristic: Lesion Location [Number; unit: participants]
  Ostial | 14 | 5 | 19
  Proximal | 91 | 42 | 133
  Mid | 100 | 56 | 156
  Distal | 19 | 22 | 41
Lesion Characteristics [Mean (Standard Deviation); unit: millimeters]
  Reference Vessel Diameter | 2.1 (0.3) | 2.2 (0.4) | 2.1 (0.3)
  Minimum Lumen Diameter | 0.6 (0.2) | 0.6 (0.2) | 0.6 (0.2)
  Lesion Length | 11.7 (5.1) | 12.9 (5.1) | 12.1 (5.1)
  Sidebranch Stenosis | 18.1 (24.6) | 16.0 (21.2) | 17.4 (23.4)
Percent Diameter Stenosis [Mean (Standard Deviation); unit: percent] | 73.5 (10.2) | 71.5 (10.4) | 72.8 (10.3)
Lesion Characteristics [Number; unit: participants] — The same participant may be included in more than one category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    Eccentric Lesion | 149 | 78 | 227
    Tortuosity, any | 20 | 23 | 43
    Calcification, any | 30 | 26 | 56
    Total Occlusion | 3 | 1 | 4
    Bifurcation | 53 | 27 | 80
    > 45 Degree Bend | 14 | 15 | 29
    > 90 Degree Bend | 0 | 0 | 0
Lesion Characteristics: American College of Cardiology (ACC)/American Heart Association (AHA) [Number; unit: participants] — Type A lesions: minimally complex, readily accessible, non angulated, smooth contour, little to no calcification, less than totally occlusive, not ostial in location, no major side branch involvement, and an absense of thrombus.
  Type B lesions: moderately complex, eccentric, moderate tortuosity and angulation, moderate or heavy calcification, total occlusion < 3 months old, ostial in location, with presence of thrombus.
  Type C lesions: severely complex, diffuse, excessive tortuosity and angulation, total occlusions > 3 months old, degenerated vein grafts and friable lesions.
  participants
    Type A | 21 | 7 | 28
    Type B1 | 73 | 21 | 94
    Type B2 | 99 | 73 | 172
    Type C | 31 | 24 | 55
Lesion Characteristic: Pre-Procedure Thrombolysis In Myocardial Infarction (TIMI) Flow [Number; unit: participants] — TIMI 0 - No perfusion TIMI 1 - Penetration with minimal perfusion TIMI 2 - Partial perfusion TIMI 3 - Complete perfusion
  participants
    TIMI 0 | 1 | 0 | 1
    TIMI 1 | 2 | 1 | 3
    TIMI 2 | 1 | 7 | 8
    TIMI 3 | 220 | 117 | 337

OUTCOME MEASURES:

1. Primary Outcome: In-stent Late Loss Measured by Quantitative Coronary Angiography (QCA)
Description: Post-procedure minimum lumen diameter (mm) minus follow-up minimum lumen diameter as determined by quantitative angiography. Minimum lumen diameter is measured within the stent at each time point.
Time Frame: 9 months post-index procedure
Population: The primary analysis population for the superiority testing of the primary endpoint, 9-month in-stent late loss, is the intent-to-treat (ITT) population, i.e. all patients who had a study device implanted at the target lesion and completed their angiographic follow-up.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | TAXUS Element | Historical Control Bare Metal Stent (BMS)
Number analyzed (Participants) | 197 | 108
millimeter | 0.38 (0.51) | 0.80 (0.53)
Statistical Analysis 1: Comparison: TAXUS Element vs Historical Control Bare Metal Stent (BMS); A superiority test of TAXUX Element vs bare metal (BMS) Express historical control. The null hypothesis that the true difference in means (TAXUS Element - BMS Express) is equal to zero was tested against the two-sided alternative that the true difference in means is different from zero. A sample size of 224 patients in the TAXUS Element group (190 after 15% attrition due to angiographic follow-up) provided 85% power; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.54 to -0.30]

2. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) at 12 Months Post-index Procedure. TLF is Defined as Any Ischemia-driven Revascularization of the Target Lesion, Myocardial Infarction (Q-wave and Non-Q-wave), or Death Related to the Target Vessel.
Description: The number of participants who experience a TLF through 365 days post-procedure out of the patients who have either had a TLF within 365 days post-procedure or who were TLF-free with last follow-up at least 335 days post-procedure.
Time Frame: 12 months post-index procedure
Population: Intent-to-Treat. All enrolled patients are included in the analysis.
Measure: Number; unit: participants
Arm/Group | TAXUS Element | Historical Control Bare Metal Stent (BMS)
Number analyzed (Participants) | 218 | 121
participants | 16 | 27
Statistical Analysis 1: Comparison: TAXUS Element vs Historical Control Bare Metal Stent (BMS); One-sided, single-sample binomial test to compare the observed TLF rate in PERSEUS SV to the pre-specified performance goal (19.5%). The normal approximation of the test statistic was used. The null hypothesis that the true TAXUS Element TLF rate is greater than or equal to the performance goal was tested against the one-sided alternative that the true rate is less than the performance goal. A sample size of 224 patients (accounting for 5% attrition to follow-up) provided 80% power; Test type: Superiority or Other; p < 0.0001, Chi-squared; 12-month TLR rate = 7.34, 95% CI 1-sided [upper limit 10.8]

ADVERSE EVENTS:
Time Frame: Serious adverse events are reported through 365 days. Non-serious adverse events exceeding 5% threshold are reported through 270 days.
Description: Per the study protocol, non-serious adverse events are reported through the 9-month follow-up assessment (primary endpoint). Past the 9-month assessment, reporting of events was limited to major adverse cardiac events and serious adverse events only.
Arm/Group | TAXUS Element | Historical Control Bare Metal Stent (BMS)
Serious Adverse Events (participants affected / at risk) | 100/224 | 70/125
Other Adverse Events (participants affected / at risk) | 75/224 | 41/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAXUS Element (N=224) | Historical Control Bare Metal Stent (BMS) (N=125)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 27 (32) | 33 (40)
Angina unstable (Cardiac disorders) | 5 (5) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 1 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 8 (8) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 12 (12) | 16 (17)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Glaucoma (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 1 (1) | 0 (0)
Implant site haematoma (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 7 (8) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac stress test abnormal (Investigations) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 2 (2) | 0 (0)
Anaemia NOS (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure NOS (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary oedema NOS (Cardiac disorders) | 0 (0) | 1 (1)
Thyroid nodule (Endocrine disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Contrast media reaction (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia NOS (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bile duct cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure NOS (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma aggravated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypertension NOS (Vascular disorders) | 0 (0) | 1 (1)
Cardiac enzymes increased (Investigations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAXUS Element (N=224) | Historical Control Bare Metal Stent (BMS) (N=125)
Angina pectoris (Cardiac disorders) | 32 (38) | 23 (24)
Nausea (Gastrointestinal disorders) | 12 (12) | 7 (8)
Non-cardiac chest pain (General disorders) | 24 (25) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 0 (0)
Catheter site haematoma (General disorders) | 5 (5) | 8 (8)
Chest pain (General disorders) | 2 (2) | 8 (10)
Fatigue (General disorders) | 9 (10) | 8 (8)

LIMITATIONS AND CAVEATS:
There were no commercially available dedicated small vessel paclitaxel-eluting stents at the time of study enrollment, thus, the PERSEUS Small Vessel comparator group does not represent the most recently available paclitaxel-eluting stents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall have the right to publish the results, provided that before publishing, the PI shall submit copies of any proposed publication or presentation to Sponsor for review at least sixty (60) days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.